CLINICAL TRIAL: NCT04720898
Title: LUNA-EMG to Enhance Lower Limb Motor Functions in Multiple Sclerosis
Brief Title: LUNA-EMG to Enhance Motor Functions in Multiple Sclerosis
Acronym: LUNA-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-372b
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LUNA-EMG (Experimental): The experimental group will receive 30 minutes of training with the LUNA-EMG once a week for 12 weeks.
  Interventions: Device: LUNA-EMG
- Control (No Intervention): The control group will receive its rehabilitation care.

INTERVENTIONS:
Device: LUNA-EMG — The LUNA-EMG (Samcom) system is a robot that allows the evaluation of muscular strength through the recording of muscle activity (electromyography - EMG) in order to provide precise objective data on the patient's muscle function. In addition to the diagnostic aspect (evaluation of muscle strength, range of motion and proprioception), the LUNA-EMG robot provides optimized range of motion's movements and a visual feedback on the patient's performance. In addition, it may enhance neuroplasticity due to the increased number of movements repetitions which could influence motor learning.
  Arms: LUNA-EMG

SUMMARY:
The aim of the present study is to evaluate the effects of training performed with the LUNA-EMG system to enhance motor functions of the lower limb in multiple sclerosis. This is a randomized open-label trial. Patients will be randomized into the intervention group (LUNA-EMG, 30-45 minutes once a week for 12 weeks) or in the control group (standard care).

The effect of the training will be measured based on the muscular strength, walking tests, proprioception and a quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* EDSS less or equal to 6.5
* Between 18 and 70 years old
* Having signed the informed consent

Exclusion Criteria:

* Acute pain syndrome
* Severe cognitive deficits
* Risk of fracture or unconsolidated fracture
* Rigid joints (spasticity, severe osteoarthritis and arthritis) or unstable joints
* Severe ataxia and apraxia
* Epilepsy
* Pacemakers and similar implants
* Insufficient skin conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Muscle strength in mV | 12 weeks
  Muscular strength is measured with a dynamometer.

SECONDARY OUTCOMES:
Timed 25-Foot Walk, seconds | 12 weeks
  The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The faster the better.
Timed Up and Go, seconds | 12 weeks
  The person must get up from the seated position and walk three meters away from the chair and then retrace their steps (turn 180 degrees) and sit down again. The faster the better.
Proprioception | 12 weeks
  Patients proprioception will be measured with the LUNA system. It calculates the distance in degree (°) between the target arm position and the arm position that the patient try to reproduce. Lower degree represent a more accurate positioning of the arm by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- CNRF, Tinlot, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No